CLINICAL TRIAL: NCT02609009
Title: Back Pain Management With Spinal Manipulation Therapy Compared to Usual Medical Care in Adolescent Idiopathic Scoliosis Patients: A Pilot Study
Brief Title: Back Pain and Spinal Manipulation in Adolescent Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Fondation Chiropratique du Québec (Other)
Responsible Party: Principal Investigator, Jean Théroux, Chiropractor, PhD student, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3928
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Back Pain; Scoliosis
Keywords: Back Pain; Adolescent Idiopathic Scoliosis; Spinal Manipulation
MeSH Terms: conditions — Back Pain; Scoliosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spinal Manipulation Therapy (Experimental): Active chiropractic care for this RCT will consist of diversified technique prone, side posture and supine manipulations with soft-tissue therapy
  Interventions: Other: Spinal Manipulation Therapy
- Usual Medical Care (Other): Control group patients will follow the usual medical visit scheduled according to their attending orthopaedists. Usual interventions generally consist in the administration of medications (NSAIDs or ibuprofen), physical therapy or exercises.
  Interventions: Other: Usual Medical Care

INTERVENTIONS:
Other: Spinal Manipulation Therapy — Intervention will consist of Diversified type adjustments. Patients will be assigned to the nearest participating chiropractic clinic and will have a complete standardized examination on their first visit. Patient will then receive a maximum of 12 treatments (3x per week for a period of 4 weeks).
  Arms: Spinal Manipulation Therapy
Other: Usual Medical Care — Usual interventions generally consist in the administration of medications (NSAIDs or ibuprofen), physical therapy or exercises. If recommended, physical therapy will be provided by the hospital physical therapy services. Physical therapy might include treatments such as massage, different electrotherapy, postural repositioning, exercises, etc
  Arms: Usual Medical Care

SUMMARY:
Adolescent idiopathic scoliosis (AIS) affects 2 - 3% of children and adolescents older than 10 years and is of unknown cause. It was initially thought that occurrences of back pain (BP) were similar to the one encounter in healthy adolescents. Recently, literature has shown that there is a two-fold prevalence of BP among AIS patients compared to healthy adolescents. As such, BP appears as a condition that might have a detrimental effect on the well-being of AIS patients and seems associated with increases in health care costs. Further, BP in adolescents would appear to be a predictive factor for adult BP. Is vertebral manipulation (VM) a viable alternative? Since 2006, four guidelines were in agreement as to the value of that approach with acute or chronic BP in adults. Unfortunately, no study was found in adolescents. The purpose of the study is to verify if VM is efficacious at improving AIS patients' back pain and to find out if it can help these patients to obtain a better quality of life and improve their spinal flexibility. Recruitment will take place at Ste Justine's hospital where patients will have 2 evaluations, conducted by an independent orthopaedist (baseline and 4 weeks). Patients will be allocated to either the experimental (VM) or the usual medical care group. Spinal manipulation treatment will last over a 4-week period. The study will be the first trial evaluating the efficacy of vertebral manipulation in adolescent idiopathic scoliosis patients with back pain. Finally, no other study was found on available and effective treatment regarding back pain management for this population. A well-structured trial is needed to provide clinicians with a better understanding and best evidence regarding treatment protocols.

DETAILED DESCRIPTION:
Introduction Adolescent Idiopathic Scoliosis (AIS) is defined by the Scoliosis Research Society (SRS) has a three-dimensional deviation of the vertebral column of unknown origin appearing in adolescents older than 10 years. Chronic non-specific back pain (CNSBP) is often associated with adolescent scoliosis patients, and the associated prevalence is almost double that of non-scoliosis healthy adolescents. Furthermore, CNSBP seems to be a predictor of CNSBP in adulthood.

Few studies evaluated BP among AIS patients and in those who did, conflicting results, regarding back pain prevalence, were observed. Among these, only two studies looked at back pain in adolescent idiopathic scoliosis. Ramirez et al. retrospectively evaluated, 2442 scoliosis adolescent patients' files establishing BP prevalence at 32%. He concluded that the established prevalence was similar to the one encountered in a general non-scoliotic adolescent population. Joncas and Labelle prospectively evaluated 239 adolescents with idiopathic scoliosis for the prevalence of BP. They observed that BP occurred in 54% of patients, and the average pain intensity was 49,4 mm. More recently, Sato's studied back pain prevalence in adolescents with idiopathic scoliosis. He conducted a large-scale cross-sectional epidemiological study, where 43 630 children aged 9 to 15-year-old were required to complete a take-home questionnaire. They reported a back pain prevalence of 58.8% in scoliosis patients compared to 32.9% in non-scoliosis patients.

Regarding BP Management in AIS Patients, a comprehensive review of the literature did not yield any study on BP management in AIS patients. Spinal manipulation therapy (SMT) is a recognised and safe treatment for low back pain and is performed primarily by chiropractors, physical therapists, and osteopaths. To the best of the investigators' knowledge, only one pilot clinical trial (Rowe 2006) has been conducted with children and adolescents diagnosed with AIS. Though under powered, results showed that SMT was associated with only minor adverse events, there was no curve progression in the treatment group, and quality of life, evaluated by the Scoliosis Quality of life Index, has not been negatively impacted.

In light of the paucity of literature on the management of back pain in nonsurgical AIS patients, and considering the lack of evidence in regards to the efficacy of SMT for back pain in adolescents, and the lack of guidance regarding management of back pain in adolescents, it would be important to evaluate the effectiveness of SMT compared to usual medical care for back pain among adolescents with idiopathic nonsurgical scoliosis.

The primary objective of this pilot study is to verify the effect of Spinal Manipulative Therapy on back pain management of adolescents with idiopathic nonsurgical scoliosis. The secondary objectives are two-fold: 1) to verify the effect of SMT on low back function, 2) to verify the feasibility and acceptability of SMT according to patients' level of satisfaction. This pilot study will be used to verify some implementation strategies before proceeding to a subsequent larger trial, such as recruitment rate, treatment compliance and loss to follow up, and adverse events.

Methods: Study Design This pilot study is a single prospective centre randomised controlled trial with one experimental and one control group. This study will be recruiting from Ste-Justine University Hospital in Montreal, Canada, and patients will be required to attend at least 80% of the treatment sessions otherwise they will be considered as non-compliant. Chiropractors will be recruited from their professional regulatory board. Different instruments will be used during this trial: questionnaires; the Brief Pain Inventory Questionnaire, and the Roland-Morris Disability Questionnaire; the modified Fingertip-to-floor distance, the modified-modified Schöber test, and the Biering-Sorenson back muscles extensor test. Patients will be evaluated upon trial entry and at 4 weeks (end of trial). Co-interventions will be documented and accounted in the analysis. Eligible patients will be randomized according to blocks of 4 to either the experimental (SMT) or the control (UMC) arm after informed consent has been obtained. The randomisation list will be generated and managed by an independent statistician. Statistical software SPSS version 22 will be used for data analyses. All analyses will be conducted under the intention-to-treat principle. To ensure balance, groups will be compared for possible confounders (age, gender, brace) at baseline. The group mean (Std. Deviation) and frequencies will be presented. Tests will be 2-tailed, and the significance level will be set at 0.05. Statistical analysis will include t-test (or Mann-Whitney) for continuous variables and χ2 for categorical variables. Considering that patient's inclusion criterion is chronic pain, and that by definition chronic pain is defined as constant over a period; the investigators expect this variable not to be time influenced. Ste-Justine University Hospital ethical committee has approved this study.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents 10 to 17-year-old of either gender
2. Both, parents and adolescents speak either English or French
3. Adolescents with a diagnosis of AIS established by one of the participating orthopaedists.
4. Pain score over 3 on scale of 0-10
5. AIS associated with mechanical back pain of at least six consecutive weeks duration with or without radiating pain to the lower extremity. Mechanical back pain is defined as pain not associated with specific identifiable aetiologies

Exclusion Criteria:

1. suffering from any metabolic, malignant or any serious organic or progressive neurological deficit.
2. any structural disturbances of the spine is present (e.g.: osteoporosis, disc herniation, spondylolisthesis, hip dysplasia and others),
3. previous back surgery for AIS
4. ongoing treatment for back pain by other health care providers
5. pregnancy
6. contraindications to SMT, other than previously mentioned, such as inflammatory or infectious conditions, blood clotting and connective tissue disorders

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2014-09; Primary Completion 2017-04-05 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Back Pain intensity | 4 weeks
  The intensity and quality of low back pain will be with the use of the Brief Pain Inventory. Questionnaire (BPI). This questionnaire is used to evaluate the quality and the intensity of pain and determine its impact upon the patient. The BPI includes 9 questions and uses an 11 -point scale (0 = "no pain"; and 10 ="pain as bad as you can imagine") to evaluate the intensity of pain at the time of being surveyed, pain at its worst, pain at rest, and average pain in the past week. This instrument also records the location of pain on a diagram using a human silhouette and requires patients to select words that best describe their pain.

SECONDARY OUTCOMES:
Physical Functioning | The RMDQ will be administered at baseline and at four week follow up.
  This outcome will be assessed by the Roland-Morris Disability Questionnaire (RMDQ).
  The RMDQ consists of 24 statements about activity limitations due to back pain, e.g. walking, lying and self-care. Patients are asked to answer yes or no to each statement. Each positive answer is worth one point with scores ranging from 0 (no disability) to 24 (severely disabled).
Spinal forward flexion | The spinal forward flexion will be administered at baseline and at four week follow up.
  Spinal forward flexion will be evaluated using the Fingertip-to-floor distance (FTFD).
  The fingertip-to-floor test is performed while the patient is standing on a platform 30 cm from the floor. The distance between the patient's third finger and the platform is measured in centimetre and assigned a positive or negative value depending if the patient is unable to reach the platform fully or if the patient reaches further than the platform.
Spinal Forward Flexion | The spinal forward flexion will be administered at baseline and at four week follow up.
  Spinal forward flexion will also be assessed using the Schöber test.
  The Schöber test uses two landmarks. An intersecting line to the line connecting both posterior superior iliac spines (PSIS) with the mid-line of the back and a mark drawn 15 cm above. Once these reference points are marked, the examiner asks the patient to bend forward as far as possible. The distance between the two-reference landmarks is then measured.
Isometric trunk extensor muscles endurance. | The spinal forward flexion will be administered at baseline and at four week follow up.
  Isometric trunk extensor muscles endurance will be evaluated using the Biering-Sorenson back muscle' extensor test. This test is performed while the patient is in a prone position with the lower half of the body below the level of the anterior superior iliac spines (ASIS) strapped to a plinth at the ankle, the knee and the hips. The test consists in measuring the amount of time a person can hold the unsupported upper body in a horizontal prone position with the lower body fixed to the examining table. The time during which the patient keeps the upper body straight and horizontal is recorded. In patients who experience no difficulty in holding the position, the test is stopped after 240 s.

CONTACTS AND LOCATIONS:
Locations (1):
- Sainte-Justine University Hospital, Montreal, Quebec, Canada